CLINICAL TRIAL: NCT03893383
Title: Knowledge- Attitude- Practice (KAP) of Post Exposure Prophylaxis for Fifth Year Dental Students of a Private Egyptian University: A Cross-sectional Study
Brief Title: Knowledge- Attitude- Practice (KAP) of Post Exposure Prophylaxis for Fifth Year Dental Students of a Private Egyptian University
Acronym: Cross-section
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar Saleem Mojahed Abou-Musallam, teacher assistant in MSA University, Cairo University
Other Study IDs: U Cairo H
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Occupational Exposure
Keywords: knowledge attitude practice questionnaire post exposure prophylaxis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
considering the increase number of occupational injuries, The aim of this study is to assess the current level of knowledge, attitude and practice of fifth year dental students as regards post exposure prophylaxis.

DETAILED DESCRIPTION:
Injuries from occupational accidents are associated with agents of biological risk, as they are the gateway to serious and potentially lethal infectious diseases. Several studies have demonstrated that dental students are among the most vulnerable to blood-borne exposure due to both their limited and restricted working area and developing skills level. This situation makes the use of post exposure prophylaxis is very important. Therefore, this study is conducting to evaluate the awareness level of fifth year dental students regarding post exposure prophylaxis.

ELIGIBILITY:
Inclusion Criteria The fifth year dental students studying at a Private Egyptian University. Dental students who agree to participate. Dental students irrespective of age and sex.

Exclusion Criteria:

• Refusal of participation from the students.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: fifth year dental students in a Private Egyptian University
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge, attitude and practice (KAP) of fifth year dental students regarding Post Exposure Prophylaxis. | one day
  the questionnaire will be given to students to be filled in one of their clinical sections

IPD SHARING:
Plan to Share IPD: Undecided